CLINICAL TRIAL: NCT01340703
Title: Vitrectomy Without Laser or Gas Tamponade for Optic Disc Pit Maculopathy
Brief Title: Vitrectomy for Optic Disc Pit Maculopathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyorin University (Other)
Responsible Party: Akito Hirakata, Kyorin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KyorinEye005
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Last update posted 2011-04-22 (Estimated); Status verified 2011-01

CONDITIONS: Optic Disc Pit Maculopathy
Keywords: optic disc pit; retinal detachment; retinoschisis; vitrectomy; posterior vitreous detachment
MeSH Terms: conditions — Retinal Detachment; Retinoschisis; Vitreous Detachment | interventions — Vitrectomy; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- optic disc pit maculopathy (Other)
  Interventions: Procedure: vitrectomy without laser or gas tamponade

INTERVENTIONS:
Procedure: vitrectomy without laser or gas tamponade — vitrectomy without laser or gas tamponade

SUMMARY:
The purpose of this study is to evaluate the efficacy of vitrectomy, without gas tamponade or laser photocoagulation to the margin of the optic nerve, for the treatment of macular detachment associated with optic disc pits and to characterize retinal manifestations during treatment of optic pit maculopathy using optical coherence tomography (OCT). Vitrectomy with induction of a PVD at the optic disc without gas tamponade or laser photocoagulation appears to be an effective method of managing macular detachment due to optic disc pits. OCT scanning pre- and postoperatively suggests that peripapillary vitreous traction with the passage of fluid into the retina through the pit is the cause of the schisis-like separation seen in optic disc pit maculopathy.

ELIGIBILITY:
Inclusion Criteria:

* eyes with optic disc pit maculopathy

Exclusion Criteria:

* eyes without macular elevation associated with optic disc pit

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2005-01; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
anatomical result | one year
  resolution of retinal detachment or retinoschisis

SECONDARY OUTCOMES:
visual acuity | one year
  preoperative and postoperative visual acuity

CONTACTS AND LOCATIONS:
Overall Officials: Akito Hirakata, MD, Principal Investigator — Kyroin University
Locations (1):
- Kyroin University Eye Center, Mitaka, Tokyo, Japan